CLINICAL TRIAL: NCT00188695
Title: A Pilot Study of MR Imaging With Ultra-small Superparamagnetic Iron Oxide for Pelvic Lymph Node Target Definition
Brief Title: Combidex USPIO - Ultra-small Superparamagnetic Iron Oxide
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Dr. Michael Milosevic, Principal Investigator, University Health Network
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-0838-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Uterine Neoplasms; Cervix Neoplasms; Bladder Neoplasms; Prostatic Neoplasms
MeSH Terms: conditions — Uterine Neoplasms; Uterine Cervical Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms | interventions — ferumoxtran-10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: MRI contrast agent Combidex (ferumoxtran-10) — Combidex as an MR-lymph node contrast agent for the detection of small lymph nodes and lymph metastases.

SUMMARY:
The purpose of this study is to test whether or not a new contrast agent called Combidex, a contrast agent formulated from ultra-small superparamagnetic iron oxide (USPIO) improves the ability of Magnetic Resonance Imaging (MRI) to see lymph nodes in the pelvis. It might also help doctors tell whether or not cancer has spread to these lymph nodes. It might allow radiotherapy to be delivered more accurately.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed endometrial, cervix, prostate (cT1-cT3) or bladder cancer
* no distant metastases
* informed consent

Exclusion Criteria:

* confirmed prostate carcinoma and PSA less than or equal to 4 or greater than 100
* radical surgery or prior cryosurgery for prostate carcinoma, previous RT, hormonal manipulation or chemotherapy
* biopsy-proven lymph node involvement
* endometrium or cervix carcinoma who have undergone recent pelvic surgery with the exclusion of D&C or biopsy
* bladder carcinoma with recent pelvic surgery with the exclusion of TURBT
* previous or concurrent cancers other than superficial basal or squamous cell skin carcinoma unless disease-free for at least 5 yrs
* contraindication to MR imaging
* hip prosthesis
* major medical or psychiatric illness
* patients with known allergy to dextran or iron-containing compounds
* patients with cirrhosis or hemochromatosis
* patients receiving another MR contrast within 2 hrs prior to the ferumoxtran-10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Improved delineation of normal pelvic lymph nodes in patients with uterine, cervical, bladder and prostate cancers. | once at time of imaging
Improved clinical target volume (CTV) definition for the purpose of adjuvant irradiation of pelvic lymph nodes using intensity modulated radiotherapy (IMRT). | once at time of imaging

SECONDARY OUTCOMES:
Comparison of target lymph node delineation between nodal imaging with USPIO and volume expansion of vascular anatomy. | once at time of imaging
Demonstration of the pattern and distribution of pelvic nodal metastases in patients with uterine, cervical, bladder and prostate cancers. | once at time of imaging

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milosevic, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada